CLINICAL TRIAL: NCT01224353
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Thioctacid Oral Tablet 600mg Once Daily in Chinese Diabetic Patients With Distal Symmetric Polyneuropathy
Brief Title: Efficacy and Safety Study of Thioctacid Oral Tablets 600mg to Treat Chinese Diabetic Patients With Distal Symmetric Polyneuropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NovaMed Pharmaceuticals Inc. (Industry)
Responsible Party: Wan Qi/Director, Neuropathic Department, Jiangsu Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM2010001
Record Dates: First submitted 2010-10-17; First posted 2010-10-20 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Diabetics
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thioctacid Oral Placebo Tablet (Placebo Comparator)
  Interventions: Other: Placebo
- Thioctacid Oral Tablet (Active Comparator)
  Interventions: Drug: lipoic acid

INTERVENTIONS:
Drug: lipoic acid — Tablet, 600mg, for oral use, 30 min before breakfast, once daily for 6 weeks
  Arms: Thioctacid Oral Tablet
Other: Placebo — Tablet, placebo, 1-week single-blind placebo treatment then, 30 min before breakfast, once daily for 6 weeks
  Arms: Thioctacid Oral Placebo Tablet

SUMMARY:
The purpose of the study is to evaluate the efficacy on overall neuropathic sensory symptom improvement of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with distal symmetric polyneuropathy (DSP).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfil all of the following criteria to be appropriate to enter into Registry (Visit 2)

  1. Provision of informed consent
  2. Females and males aged from 18 to 75 (inclusive), who were definitely diagnosed with diabetes
  3. HbA1C< 10％
  4. Moderate neuropathy according to Neuropathy Disability Score (NDS) >= 4 points. Difference in score between left and right foot is not to be higher than 2 points
  5. Total Symptom Score (TSS) > 6.5 points
  6. At least one of the four symptoms of the TSS has occurred continuously over the last 3 months before screening
  7. Other concomitant treatments (the drugs and their dosage) have been stable over 1 month before screening Subjects must fulfil all of the following criteria before randomization：
  8. TSS > 5 points
  9. TSS range (maximum TSS - minimum TSS during Run-in Period) < 3 points during the Run-in Period
  10. Compliance in Run-in Period > 85%

Exclusion Criteria:

1. Neurologic disease other than diabetic neuropathy that may produce weakness, sensory loss, or autonomic symptoms or test abnormality
2. Peripheral vascular disease severe enough to cause intermittent claudication or ischemic ulcers
3. Patients who have been hospitalized due to glucopenia or ketoacidosis in the last 3 month
4. Present ulcers on lower limbs of any cause
5. Antioxidant therapy within the last 1 month before screening (Vitamin E> 400IU, Vitamin C> 200mg once daily for continuous 2 weeks)
6. Any ALA therapy within the last1 month before screening
7. Opioid analgesic therapy within the last 1 month before screening
8. History of mental, psychological or behavioral conditions rendering the patient unable to follow the protocol
9. History of malignant tumors in the past 5 years except for basal cell carcinoma
10. Any severe systematic diseases, at the investigator's discretion, which will make it undesirable for the patient to participate in the trial or which could jeopardize compliance with the trial protocol,
11. ALT or AST > 2.5 ´ upper limit of reference range
12. Cr > 1.8mg/dL ( > 159µmol/L) for males or > 1.6mg/dL ( > 141µmol/L) for females
13. History of hypersensitive to the active ingredients or excipients of ALA
14. Participation in a clinical study or treatment with a non-approved experimental medication in the last 1 month
15. Pregnant or breast-feeding women, or women of childbearing age without appropriate contraception measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy on overall neuropathic sensory symptom improvement of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with distal symmetric polyneuropathy (DSP) | 6 weeks
  Changes from baseline in Total Symptom Score (TSS) from week 1 to week 6 will be computed and summarized in an Area Under the Curve (AUC).

SECONDARY OUTCOMES:
To evaluate each sensory symptom improvement of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with DSP | 6 weeks
  Changes in the individual symptom scores of the TSS (Stabbing pain, burning, paraesthesia, numbness)
To evaluate onset time of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with DSP | 6 weeks
To evaluate response rate of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with DSP | 6 weeks
To evaluate the tolerability and safety of Thioctacid tablet 600mg once daily vs. placebo in 6-weeks' treatment in Chinese diabetic patients with DSP | 6 weeks
  Number of adverse events and standard laboratory tests will be the Measures of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Qi Wan, Principal Investigator — Jiangsu Provincial People's Hospital
Locations (5):
- China (5):
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu